CLINICAL TRIAL: NCT07082686
Title: A Single-arm, Multi-center, Open-label, Phase 2 Study to Evaluate the Efficacy and Safety of ICP-248 in Subjects With Relapsed or Refractory Mantle Cell Lymphoma
Brief Title: A Study to Evaluate the Efficacy and Safety of ICP-248 in Subjects With Relapsed or Refractory Mantle Cell Lymphoma (APEX-06)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICP-CL-01206
Record Dates: First submitted 2025-07-15; First posted 2025-07-24 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-08

CONDITIONS: Relapsed or Refractory Mantle Cell Lymphoma (MCL)
MeSH Terms: conditions — Recurrence; Lymphoma, Mantle-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICP-248Tablets (Experimental)
  Interventions: Drug: ICP-248

INTERVENTIONS:
Drug: ICP-248 — Eligible patients will receive ICP-248 orally as per the protocol

SUMMARY:
This is a single-arm, multi-center, open-label, phase 2 study to evaluate the efficacy and safety of ICP-248 in subjects with relapsed or refractory mantle cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old.
* Histopathologically confirmed MCL expressing Cyclin D1 and/or t (11;14) chromosomal translocation.Formalin-fixed paraffin-embedded (FFPE) tissues or sections for diagnosis must be provided. It is for the approval of pathological diagnosis by the central pathology laboratory.
* The patient was diagnosed with relapsed or refractory mantle cell lymphoma, and the previous treatment needs to meet the following requirements:

  * Failure of at least one adequate prior line of anti-CD20-containing therapy;
  * Failure of at least one adequate prior line of BTK inhibitor (BTKi)-containing therapy.
* Failure of the last line of therapy.
* At least one measurable lesion according to the Lugano 2014 criteria,.
* ECOG performance status of 0-2 .

Exclusion Criteria

* Blastoid or pleomorphic mantle cell lymphoma (MCL).
* Current or prior history of central nervous system (CNS) lymphoma.
* Prior use of BCL-2 inhibitors (e.g., venetoclax/ABT-199, etc.).
* Autologous stem cell transplantation or cellular therapy within 3 months prior to the first dose of ICP-248.
* Prior allogeneic hematopoietic stem cell transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-08-21 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) according to Lugano 2014 assessed by the independent review committee (IRC) | 3 years

SECONDARY OUTCOMES:
According to Lugano 2014: IRC and investigator assessed complete response rate (CRR) | 3 years
Investigator-assessed ORR | 3 years
According to Lugano 2014: IRC and investigator assessed disease control rate (DCR). | 3 years
According to Lugano 2014: IRC and investigator assessed duration of response (DOR). | 3 years
According to Lugano 2014: IRC and investigator assessed time to initial response (TTR). | 3 years
According to Lugano 2014: IRC and investigator assessed progression-free survival (PFS) . | 3 years
Overall survival (OS) | 3 years
Adverse event (AE) assessed according to CTCAE v5.0 criteria | 3 years
Functional Assessment Of Cancer Therapy-Lymphoma (Fact-Lym) and European Quality Of Life Five Dimension Five Level Scale Questionnaire (Eq-5D-5L). | 3 years
Area under the plasma concentration versus time curve (AUC) | 3 years
minimal residual disease （MRD） status | 3 years
Peak Plasma Concentration (Cmax) | 3 years
Time of maximum observed plasma(Tmax) | 3 years
Trough concentration(Ctrough) | 3 years
Apparent clearance (CL/F) | 3 years

CONTACTS AND LOCATIONS:
Locations (29):
- China (29):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - West China Hospital of Sichuan University, Chengdu, Chengdu
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First Affiliated Hospital of University of South China, Hengyang, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shandong Provincial Hospital Affiliated to Shandong First Medical University, Jinan, Shandong
  - Shandong Cancer Hospital, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xian, Shanxi
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - The Second People's Hospital of Yibin, Yibin, Sichuan
  - Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - The Affiliated Cancer Hospital of Xinjiang Medical University, Xinjiang, Xinjiang
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang